CLINICAL TRIAL: NCT00493337
Title: A Community Pharmacist-led Intervention to Improve Adherence to Lipid-lowering Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utrecht Institute for Pharmaceutical Sciences (Other)
Collaborators: Service Apotheek BV (Unknown); Harvard University (Other); Department of Clinical Pharmacy, University Medical Centre St Radboud, The Netherlands. (Other); Scientific Institute for Dutch Pharmacists, The Netherlands (Other); Federation of Patients and Consumer Organisations in the Netherlands (Unknown)
Responsible Party: BLG van WIjk, Utrecht Institute for Pharmaceutical Sciences, Utrecht University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NL18496.041.07
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2007-06

CONDITIONS: Hypercholesterolemia
Keywords: Adherence; Compliance; Statins; Intervention; Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention)
- Advanced counseling (Experimental)
  Interventions: Behavioral: advanced adherence counseling+reminder
- Compliance Card only (Active Comparator)
  Interventions: Device: Compliance Card

INTERVENTIONS:
Behavioral: advanced adherence counseling+reminder
  Arms: Advanced counseling
Device: Compliance Card
  Arms: Compliance Card only

SUMMARY:
The objective of the study is to test the effectiveness of a community pharmacist-led intervention to increase adherence to lipid lowering treatment.

DETAILED DESCRIPTION:
Medication non-adherence represents an important threat to the health of the Western people. A large number of pharmacy records based studies demonstrated that adherence to lipid lowering treatment in daily practice is substantially worse compared to adherence observed in the controlled setting of randomized controlled trials. In addition, the relationship between non-adherence with statin-treatment assessed with pharmacy records and cardiovascular outcomes has been convincingly demonstrated. This implies that pharmacy records can and should be used to identify non-adherent patients and thus patients at risk for major cardiovascular events. Using this data, community pharmacists can play a more substantive role in developing the concept of pharmaceutical care. The objective of the study is to test the effectiveness of a community pharmacist-led intervention to increase adherence to lipid lowering treatment.

ELIGIBILITY:
Inclusion Criteria:

* Suboptimal adherent to statin treatment
* Older than 65 years
* Responsible for own medication intake

Exclusion Criteria:

* Life expectancy shorter than 6 months
* Institutionalized
* User of medication blisters

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 373 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be mean differences in adherence over 365 days after randomization by comparing the two intervention groups with the control group. | one year

SECONDARY OUTCOMES:
Mean differences in adherence over 180 days after randomization by comparing the two intervention groups with the control group. | 180 days
Mean differences in adherence over 270 days after randomization by comparing the two intervention groups with the control group. | 270 days
If the pre-specified effect on mean adherence is measured, change in LDL-C will also be assessed. | 365 days
Complete discontinuation defined as more than 182 consecutive days of the one year observation period uncovered (<50%). | one year

CONTACTS AND LOCATIONS:
Overall Officials: Boris LG Van Wijk, PharmD, PhD, Principal Investigator — Department of Pharmacoepidemiology & Pharmacotherapy, Utrecht Institute for Pharmaceutical Sciences, Utrecht University; Anthonius De Boer, MD, PhD, Study Director — Department of Pharmacoepidemiology & Pharmacotherapy, Utrecht Institute for Pharmaceutical Sciences, Utrecht University; Olaf H Klungel, PharmD, PhD, Study Chair — Department of Pharmacoepidemiology & Pharmacotherapy, Utrecht Institute for Pharmaceutical Sciences, Utrecht University; William H Shrank, MD, MSHS, Study Chair — Division of Pharmacoepidemiology and Pharmacoeconomics, Department of Medicine, Brigham and Women's Hospital and Harvard Medical School, Boston; Peter AG De Smet, PharmD, PhD, Study Chair — Scientific Institute of Dutch Pharmacists, The Hague; Eibert R Heerdink, PhD, Study Chair — Department of Pharmacoepidemiology & Pharmacotherapy, Utrecht Institute for Pharmaceutical Sciences, Utrecht University; Emma Giesen, PharmD, Study Chair — Service Apotheek BV; Marnix Westein, PharmD, Study Chair — Federation of Patients and Consumer Organisations in the Netherlands, Utrecht, The Netherlands; Martina Teichert, PharmD, Study Chair — Scientific Institute of Dutch Pharmacists, The Hague, The Netherlands
Locations (1):
- Service Apotheek BV, Enter, Netherlands